CLINICAL TRIAL: NCT02799836
Title: The Effect of Light Deprivation on Visual Functions in Adult Amblyopes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study never started, did not receive IRB approval and was closed administratively at the site. Therefore, no subjects were recruited or enrolled.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Melanie Kazlas, PI, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00008306
Record Dates: First submitted 2016-02-18; First posted 2016-06-15 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Amblyopia; Anisometropia; Visual Impairment
MeSH Terms: conditions — Amblyopia; Anisometropia; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Light deprived study subjects (Experimental): Study subjects who are blindfolded for 48 hours
  Interventions: Device: Blindfold

INTERVENTIONS:
Device: Blindfold — Study subjects will be blindfolded to create an environment of complete light deprivation which will be worn for 48 hours.

SUMMARY:
Amblyopia is a significant health problem, affecting up to 4% of the population in the United States. Amblyopia, commonly known as "lazy eye," is a developmental visual disorder in which one or both eyes suffer from poor vision as a result of being disadvantaged in early life. Strabismus, or eye misalignment, such as crossed eyes (esotropia) or wandering eyes (exotropia), and anisometropia, or a power difference between the eyes, are the most common causes of amblyopia. If conventional treatment, such as patching the better seeing eye, is not initiated during the critical period of visual development, lasting visual impairment may persist throughout life. This critical period of visual development has been thought to end around age 10. However, recent research has demonstrated that the critical period of visual development can be extended into adulthood. Complete light deprivation in animal models has restored plasticity in the visual cortex and has demonstrated drastic recovery of vision in amblyopic eyes. The objective of this pilot study is to evaluate the impact of complete light deprivation on visual function in a cohort of human adults with severe amblyopia from anisometropia.

ELIGIBILITY:
Inclusion Criteria:

* Amblyopia, defined as decreased vision, less than or equal to 20/100, in one eye secondary to anisometropia
* Age 18-50 years

Exclusion Criteria:

* Strabismus
* Eye pathology, such as cataract, corneal disorder, maculopathy, glaucoma,
* Mental health diagnosis, such as depression, schizophrenia, bipolar disorder or anxiety disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Logmar visual acuity | Measured at 60 minutes after blindfold is removed
Logmar visual acuity | Measured at one week after blindfold is removed

IPD SHARING:
Plan to Share IPD: Yes
Study subject's visual acuity before and after the intervention will be given to the study subject.